CLINICAL TRIAL: NCT05253274
Title: The Effect of Virtual Reality Glasses Applied During Emergency Surgical Intervention With Local Anesthesia on Patients Anxiety
Brief Title: The Effect of Virtual Reality Glasses Applied During Emergency Surgical Intervention
Acronym: Virtual
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Merve TOPAL, Nurse, Mersin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MersinUn
Record Dates: First submitted 2022-02-06; First posted 2022-02-23 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Anxiety
Keywords: Anxiety; Virtual reality glasses; Emergency Surgery
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: prospective, parallel, two arm, randomized controlled clinical trial
Masking Description: The researchers will involve in the data analysis and statistics stages will blind to the group assignment. Patients in study can not be blinded. Also, the person who performed the measurements cannot be blinded due to the nature of VR application. A statistician will analyze the data, and the findings will be reported.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality application group (Experimental): VR application will be applied to the experimental group during the emergency surgical intervention under local anesthesia.
  Interventions: Device: Virtual Reality Glasses
- Control (No Intervention): The patients in the control group routinely receives standard care in the emergency service. No application will be made to the control group.

INTERVENTIONS:
Device: Virtual Reality Glasses — In addition to the routine practice of the emergency service, the virtual reality (VR) group will watch a video with VR glasses during the emergency surgical intervention under local anesthesia. Before the emergency surgery, the patients will be asked to wear a VR glasses compatible with mobile phones with android operating system and a headset that minimizes sound loss. Patients will be shown their preferred 3D licensed video software with relaxing music in the background. VR glasses will be put on the patients before starting the emergency surgical procedure under local anesthesia and applied until the procedure was completed. Patients will be asked to refill the The State Anxiety Inventory at the end of the emergency surgical intervention. At the same time, blood pressure, heart rate, respiratory rate, SpO2 values will be monitored on a portable monitor.
  Arms: Virtual Reality application group

SUMMARY:
This randomized controlled trial evaluates the effect of virtual reality glasses applied during emergency surgical intervention with local anesthesia on patients anxiety. This study hypothesizes that virtual reality glasses reduces anxiety.

DETAILED DESCRIPTION:
The sample of this study consisted of 138 patients in the experimental (n=69) and control groups (n=69). Virtual Reality (VR) application will be applied to the experimental group during the emergency surgical intervention under local anesthesia. Anxiety level will be assessed with the Spielberger State Anxiety Scale and measured by physiological responses of anxiety such as systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR), respiratory rate (RR) and peripheral oxygen saturation (SpO2) before and after VR application. In the control group, no application will be made except for standard care only.

ELIGIBILITY:
Inclusion Criteria:

* Emergency surgical intervention with local anesthesia,
* Between the ages of 18-65,
* Conscious, oriented and cooperative,
* Able to read and understand Turkish,
* Agree to participate in the study
* Does not have physical problems that will prevent the application of virtual reality glasses,
* No previous experience with virtual reality glasses,
* Not diagnosed with anxiety,
* Does not use drugs for anxiety,
* Does not use alcohol and/or drugs,
* No mental illness
* Patients who signed the Informed Consent Form/Written Consent Form

Exclusion Criteria:

* No emergency surgical intervention with local anesthesia,
* Those under the age of 18, over the age of 65,
* Unconscious, oriented and uncooperative,
* Can't read and understand Turkish,
* Those who do not agree to participate in the study,
* Having a physical problem that will prevent the application of virtual reality glasses,
* Diagnosed with anxiety,
* Using drugs for anxiety (anxiolytic, antidepressant, antipsychotic, etc.),
* Using alcohol and/or drugs,
* Having a mental disorder,
* Patients who did not sign the Informed Consent Form/Written Consent Form

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
Anxiety evaluated using the State Anxiety Scale | Change from baseline and ten minutes
  Scores ranging from 20 to 80 points are obtained in the scale. In the total score obtained from the scale in scoring the scale, 0-19 points indicate the absence of anxiety, 20-39 points indicate mild anxiety, 40-59 points indicate moderate anxiety, and 60-79 points indicate severe anxiety level. Higher state anxiety scores indicate that anxiety level is also high.

SECONDARY OUTCOMES:
Change systolic blood pressure | During emergency surgery with Local Anesthesia
  Determine patients physiological responses to anxiety (systolic blood pressure) before and after virtual reality application The researchers will measure the systolic blood pressure of the patients in the control group before and after emergency surgery with local anesthesia, and before and after the application to the experimental group after the virtual reality application. At the same time, systolic blood pressure values will be monitored on a portable monitor (8000c, Shenzhen Comen Medical Instruments Co., Ltd., China).
Change diastolic blood pressure | During emergency surgery with Local Anesthesia
  Determine patients' physiological responses to anxiety (diastolic blood pressure) before and after virtual reality application The researchers will measure the diastolic blood pressure of the patients in the control group before and after emergency surgery with local anesthesia, and before and after the application to the experimental group after the virtual reality application. At the same time, diastolic blood pressure values will be monitored on a portable monitor (8000c, Shenzhen Comen Medical Instruments Co., Ltd., China).
Change heart rate | During emergency surgery with Local Anesthesia
  Determine patients' physiological responses to anxiety (heart rate) before and after virtual reality application The researchers will measure heart rate of the patients in the control group before and after emergency surgery with local anesthesia, and before and after the application to the experimental group after the virtual reality application. At the same time, heart rate values will be monitored on a portable monitor (8000c, Shenzhen Comen Medical Instruments Co., Ltd., China).
Change respiratory rate | During emergency surgery with Local Anesthesia
  Determine patients' physiological responses to anxiety (respiratory rate) before and after virtual reality application The researchers will measure respiratory rate of the patients in the control group before and after emergency surgery with local anesthesia, and before and after the application to the experimental group after the virtual reality application. At the same time, respiratory rate values will be monitored on a portable monitor (8000c, Shenzhen Comen Medical Instruments Co., Ltd., China).
Change peripheral oxygen saturation | During emergency surgery with Local Anesthesia
  Determine patients' physiological responses to anxiety (peripheral oxygen saturation) before and after virtual reality application The researchers will measure peripheral oxygen saturation of the patients in the control group before and after emergency surgery with local anesthesia, and before and after the application to the experimental group after the virtual reality application. At the same time, peripheral oxygen saturation values will be monitored on a portable monitor (8000c, Shenzhen Comen Medical Instruments Co., Ltd., China).

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Altun Ugras, Doctorate, Study Director — Mersin University
Locations (1):
- Turkey, Mersin University,, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gong M, Dong H, Tang Y, Huang W, Lu F. Effects of aromatherapy on anxiety: A meta-analysis of randomized controlled trials. J Affect Disord. 2020 Sep 1;274:1028-1040. doi: 10.1016/j.jad.2020.05.118. Epub 2020 May 26. PMID 32663929